CLINICAL TRIAL: NCT02727036
Title: Effect of Supplementation With Pumpkin Seed Oil Versus Pumpkin Seeds on Blood Pressure and Menopausal Symptoms in Non-hypertensive Postmenopausal Women
Brief Title: Effect of Pumpkin Seed Oil or Pumpkin Seeds on Blood Pressure and Menopausal Symptoms in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17696
Record Dates: First submitted 2016-03-21; First posted 2016-04-04 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Hypertension; Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pumpkin seed oil (Experimental): Pumpkin seed oil (1g) capsules - 2 capsules per day for 12 weeks
  Interventions: Dietary Supplement: Pumpkin seed oil
- Pumpkin seeds (Active Comparator): Packet of pumpkin seeds (4.1 grams /~0.15ounces) - 1 pack per day for 12 weeks
  Interventions: Dietary Supplement: Pumpkin seeds

INTERVENTIONS:
Dietary Supplement: Pumpkin seed oil — 1 gram capsule of Pumpkin seed oil.
  Arms: Pumpkin seed oil
Dietary Supplement: Pumpkin seeds — 4.1 grams (1½ teaspoons/~0.15ounces) of pumpkin seeds
  Arms: Pumpkin seeds

SUMMARY:
The purpose of this randomized control trial is to compare the effect of pumpkin seed oil 2g/day with pumpkin seeds given as a dose of 1½ teaspoons/ 4.1 grams a day to provide 2g of lipid (equivalent to 2 grams of oil) on BP (systolic and diastolic), endothelial function, serum lipids, C-reactive protein (CRP) concentrations, and menopausal symptoms in postmenopausal women.

DETAILED DESCRIPTION:
At the onset of menopause CVD rates increase in women. A beneficial effect of pumpkin seed oil on blood pressure has been observed in postmenopausal women. More than 1 in 3 female adults have some form of cardiovascular disease (CVD), which is affected by blood pressure.

Pumpkin seed is a good source of phytoestrogens. Phytoestrogens are compounds found in plants and are comparable to human estrogen, capable of producing estrogenic effects. Studies in post menopausal women have demonstrated that pumpkin seed oil, at a dose of 2g per day for 12 weeks can decrease blood pressure and reduce menopausal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Non-hypertensive with blood pressure less than140/90 mmHg
* Post menopausal women or had a bilateral oophorectomy

Exclusion Criteria:

* Hypotensive women with BP <90/60
* Taking medications to manage blood pressure and blood lipids
* Taking estrogen supplements or on hormone replacement therapy
* Taking pumpkin seed oil supplements
* Consuming pumpkin seeds more than ¼ cup a month
* Diagnosed with depression and taking antidepressants

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure | change measured - baseline and 12 weeks

SECONDARY OUTCOMES:
Change in Total Cholesterol level (mg/dl) | change measured - baseline and 12 weeks
Change in Plasma Triglycerides (mg/dl) | change measured - baseline and 12 weeks
Change in Plasma High-Density Lipoprotein Cholesterol (mg/dl) | change measured - baseline and 12 weeks
  High-density Lipoprotein-C
Change in Plasma Low-Density Lipoprotein Cholesterol (mg/dl) | change measured - baseline and 12 weeks
Change in C-reactive protein (CRP) | change measured - baseline and 12 weeks
Change in Endothelial Function | change measured - baseline and 12 weeks
  Endothelial function will be assessed using a computer based non-invasive peripheral arterial tonometer (Endo-PAT 2000, Itamar Medical Ltd.).

CONTACTS AND LOCATIONS:
Overall Officials: Madhura Maiya, MS, Principal Investigator — Texas Woman's University; Carolyn Moore, PhD, Study Chair — Texas Woman's University
Locations (1):
- Texas Woman's University, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gossell-Williams M, Lyttle K, Clarke T, Gardner M, Simon O. Supplementation with pumpkin seed oil improves plasma lipid profile and cardiovascular outcomes of female non-ovariectomized and ovariectomized Sprague-Dawley rats. Phytother Res. 2008 Jul;22(7):873-7. doi: 10.1002/ptr.2381. PMID 18567058
- [Result] Gossell-Williams M, Hyde C, Hunter T, Simms-Stewart D, Fletcher H, McGrowder D, Walters CA. Improvement in HDL cholesterol in postmenopausal women supplemented with pumpkin seed oil: pilot study. Climacteric. 2011 Oct;14(5):558-64. doi: 10.3109/13697137.2011.563882. Epub 2011 May 5. PMID 21545273